CLINICAL TRIAL: NCT02190604
Title: A Randomized, Double Blind Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Pharmacodynamics of Single and Multiple Ascending Doses of QBW251 in Healthy Subjects and Multiple Doses in Cystic Fibrosis Patients
Brief Title: Safety, Tolerability, Pharmacokinetics, and Preliminary Pharmacodynamics of QBW251 in Healthy Subjects and Cystic Fibrosis Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQBW251X2101; 2011-005085-37 (EudraCT Number)
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2019-03

CONDITIONS: Cystic Fibrosis
Keywords: FEV1- Forced Expiratory volume; LCI - Lung Clearance Index; CFTR - cystic fibrosis transmembrane conductance regulator; cystic fibrosis; allergic bronchopulmonary aspergillosis
MeSH Terms: conditions — Cystic Fibrosis; Aspergillosis, Allergic Bronchopulmonary | interventions — icenticaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (20):
- Part 1 Cohort 1: QBW251 (Experimental): Single dose of QBW251 10 mg in Healthy Volunteers. Each treatment period was comprised of a baseline period (Day -1), an inpatient dosing period (Days 1 to 3), three follow-up visits (Days 4, 5, and 8), and one end-of-treatment-period evaluation performed 14 days after the dose of study drug (Day 15).
  Interventions: Drug: QBW251
- Part 1 Cohort 2: QBW251 (Experimental): Single dose of QBW251 25 mg in Healthy Volunteers. Each treatment period was comprised of a baseline period (Day -1), an inpatient dosing period (Days 1 to 3), three follow-up visits (Days 4, 5, and 8), and one end-of-treatment-period evaluation performed 14 days after the dose of study drug (Day 15).
  Interventions: Drug: QBW251
- Part 1 Cohort 3: QBW251 (Experimental): Single dose of QBW251 75 mg in Healthy Volunteers. Each treatment period was comprised of a baseline period (Day -1), an inpatient dosing period (Days 1 to 3), three follow-up visits (Days 4, 5, and 8), and one end-of-treatment-period evaluation performed 14 days after the dose of study drug (Day 15).
  Interventions: Drug: QBW251
- Part 1 Cohort 4: QBW251 (Experimental): Single dose of QBW251 150 mg in Healthy Volunteers. Each treatment period was comprised of a baseline period (Day -1), an inpatient dosing period (Days 1 to 3), three follow-up visits (Days 4, 5, and 8), and one end-of-treatment-period evaluation performed 14 days after the dose of study drug (Day 15).
  Interventions: Drug: QBW251
- Part 1 Cohort 5: QBW251 (Experimental): Single dose of QBW251 300 mg in healthy volunteers. Each treatment period was comprised of a baseline period (Day -1), an inpatient dosing period (Days 1 to 3), three follow-up visits (Days 4, 5, and 8), and one end-of-treatment-period evaluation performed 14 days after the dose of study drug (Day 15).
  Interventions: Drug: QBW251
- Part 1 Cohort 6: QBW251 (Experimental): Single dose of QBW251 500 mg in Healthy Volunteers. Each treatment period was comprised of a baseline period (Day -1), an inpatient dosing period (Days 1 to 3), three follow-up visits (Days 4, 5, and 8), and one end-of-treatment-period evaluation performed 14 days after the dose of study drug (Day 15).
  Interventions: Drug: QBW251
- Part 1 Cohort 6: QBW251(fed) (Experimental): Single dose of QBW251 500 mg (fed). single dose with food for a preliminary assessment of the effect of food on the absorption of QBW251 in Healthy Volunteers. Each treatment period was comprised of a baseline period (Day -1), an inpatient dosing period (Days 1 to 3), three follow-up visits (Days 4, 5, and 8), and one end-of-treatment-period evaluation performed 14 days after the dose of study drug (Day 15).
  Interventions: Drug: QBW251
- Part 1 Cohort 7: QBW251 (Experimental): Single dose of QBW251 750 mg in Healthy Volunteers. Each treatment period was comprised of a baseline period (Day -1), an inpatient dosing period (Days 1 to 3), three follow-up visits (Days 4, 5, and 8), and one end-of-treatment-period evaluation performed 14 days after the dose of study drug (Day 15).
  Interventions: Drug: QBW251
- Part 1 Cohort 8: QBW251 (Experimental): Single dose of QBW251 1000 mg in Healthy Volunteers. Each treatment period was comprised of a baseline period (Day -1), an inpatient dosing period (Days 1 to 3), three follow-up visits (Days 4, 5, and 8), and one end-of-treatment-period evaluation performed 14 days after the dose of study drug (Day 15).
  Interventions: Drug: QBW251
- Part 1 Placebo (Placebo Comparator): Placebo to QBW251 in all cohorts of part 1 in Healthy Volunteers. Each treatment period was comprised of a baseline period (Day -1), an inpatient dosing period (Days 1 to 3), three follow-up visits (Days 4, 5, and 8), and one end-of-treatment-period evaluation performed 14 days after the dose of study drug (Day 15).
  Interventions: Drug: Placebo
- Part 2 Cohort 1: QBW251 (Experimental): Multiple doses of QBW25 150 mg qd in Healthy Volunteers. 14-day treatment period, follow-up study visits (Days 18, 22 and 29) and one End-of-Study evaluation (Day 36).
  Interventions: Drug: QBW251
- Part 2 Cohort 2: QBW251 (Experimental): Multiple doses of QBW251 400 mg qd in Healthy Volunteers. 14-day treatment period, follow-up study visits (Days 18, 22 and 29) and one End-of-Study evaluation (Day 36).
  Interventions: Drug: QBW251
- Part 2 Cohort 3: QBW251 (Experimental): Multiple doses of QBW251 750 mg qd in Healthy Volunteers. 14-day treatment period, follow-up study visits (Days 18, 22 and 29) and one End-of-Study evaluation (Day 36).
  Interventions: Drug: QBW251
- Part 2 Cohort 4: QBW251 (Experimental): Multiple doses of QBW251 450 mg bid in Healthy Volunteers. 14-day treatment period, follow-up study visits (Days 18, 22 and 29) and one End-of-Study evaluation (Day 36).
  Interventions: Drug: QBW251
- Part 2 Cohort 5: QBW251 (Experimental): Multiple doses of QBW251 750 mg bid in Healthy Volunteers. 14-day treatment period, follow-up study visits (Days 18, 22 and 29) and one End-of-Study evaluation (Day 36).
  Interventions: Drug: QBW251
- Part 2 Placebo (Placebo Comparator): Placebo to QBW251 in all cohorts of part 2 in Healthy Volunteers. 14-day treatment period, follow-up study visits (Days 18, 22 and 29) and one End-of-Study evaluation (Day 36).
  Interventions: Drug: Placebo
- Part 3 Cohort 1: QBW251 (Experimental): 150 mg b.i.d. Multiple doses. Patients having a class III, IV, V, or VI mutation on one allele and any other CFTR mutation on the other allele in patients. treatment period (Day 1 to Day 14) with study visits on Days 1, 4, 7 and 14 with follow-up visits on Days 15, 28 and 42.
  Interventions: Drug: QBW251
- Part 3 Cohort 2: QBW251 (Experimental): 450 mg b.i.d. Multiple doses. Patients having a class III, IV, V, or VI mutation on one allele and any other CFTR mutation on the other allele in patients. treatment period (Day 1 to Day 14) with study visits on Days 1, 4, 7 and 14 with follow-up visits on Days 15, 28 and 42.
  Interventions: Drug: QBW251
- Part 3 Cohort 3: QBW251 (Experimental): 450 mg b.i.d. Multiple doses. Patients who are homozygous for the F508del mutation in patients. treatment period (Day 1 to Day 14) with study visits on Days 1, 4, 7 and 14 with follow-up visits on Days 15, 28 and 42.
  Interventions: Drug: QBW251
- Part 3 Placebo (Placebo Comparator): Placebo to QBW251 in all cohorts of part 3 in patients. treatment period (Day 1 to Day 14) with study visits on Days 1, 4, 7 and 14 with follow-up visits on Days 15, 28 and 42.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Capsule- oral dose
  Arms: Part 1 Placebo; Part 2 Placebo; Part 3 Placebo
Drug: QBW251 — Capsule - oral dose
  Arms: Part 1 Cohort 1: QBW251; Part 1 Cohort 2: QBW251; Part 1 Cohort 3: QBW251; Part 1 Cohort 4: QBW251; Part 1 Cohort 5: QBW251; Part 1 Cohort 6: QBW251; Part 1 Cohort 6: QBW251(fed); Part 1 Cohort 7: QBW251; Part 1 Cohort 8: QBW251; Part 2 Cohort 1: QBW251; Part 2 Cohort 2: QBW251; Part 2 Cohort 3: QBW251; Part 2 Cohort 4: QBW251; Part 2 Cohort 5: QBW251; Part 3 Cohort 1: QBW251; Part 3 Cohort 2: QBW251; Part 3 Cohort 3: QBW251

SUMMARY:
This study is designed to assess the safety, tolerability, pharmacokinetics and preliminary pharmacodynamics (proof of concept) of QBW251 in healthy subjects and cystic fibrosis patients following single and multiple doses. This first-in-human and proof of concept study will consist of 4 parts, with Parts 1 and 2 in healthy volunteers and Parts 3 and 4 in cystic fibrosis patients.

ELIGIBILITY:
Key inclusion criteria (Parts 1 and 2)

* Healthy female (of non-childbearing potential) and male subjects of 18 to 55 years of age (inclusive)
* Body mass index (BMI) must be within the range of 15 to 30 kg/m2
* Oxygen saturation (O2) at screening must be ≥ 96% on room air.

Key exclusion criteria (Parts 1 and 2)

* Use of any prescription drugs or herbal supplements within four (4) weeks prior to dosing or within 5 half-lives of the drug, whichever is longer
* Over-the-counter (OTC) medication (including vitamins, dietary supplements) within two (2) weeks prior to dosing
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
* Unwilling to avoid direct sun exposure by covering exposed skin, using topical sun block and wearing sunglasses from the first dose of study drug to the end of participation in the study
* Pregnant or nursing (lactating) women.

Key inclusion criteria (Parts 3 and 4):

* Male and female patients of 18 to 65 years of age (inclusive) with a confirmed diagnosis of cystic fibrosis as per the Cystic Fibrosis Foundation (CFF) consensus guidelines
* Heterozygous with one allele represented as any CFTR mutation and the other allele must represent a class III, IV, V, VI CFTR mutation (Note: since the CFTR mutation, F508del, can be considered either a class II or III mutation, heterozygous CF patients that have one allele that contains F508del, must have the other allele contain a class III (i.e., not F508del), IV, V, or VI mutation). Patients with F508del/F508del mutation should only be included in Part 3 Cohort 3.
* Body mass index (BMI) must be within the range of 15-35 kg/m2
* FEV1 at Screening must be 40 to 100% predicted (inclusive) by NHANES/Hankinson standards
* Oxygen saturation (O2) at screening must be > 90% on room air.

Key exclusion criteria (Parts 3 and 4)

* Use of herbal supplements within four (4) weeks prior to dosing or within 5 half-lives of the supplement, whichever is longer
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
* Unwilling to avoid direct sun exposure by covering exposed skin, using topical sun block and wearing sunglasses from the first dose of study drug to the end of participation in the study
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, UNLESS they are using highly effective contraception
* Any changes in concomitant medications for 14 days prior to screening
* History or clinical evidence of pancreatic injury or pancreatitis; clinical evidence of liver disease or liver injury as indicated by clinically significant abnormal liver function tests as judged by the investigator such as SGOT, SGPT, GGT, alkaline phosphatase, or serum bilirubin
* History or presence of impaired renal function as indicated by abnormal creatinine or BUN values or abnormal urinary constituents (e.g., albuminuria)
* History of Burkholderia cepacia respiratory tract infection (must have at least two negative cultures and no positive cultures in the past 18 months prior to screening to be eligible for enrollment)
* Sexually active males unless they use a condom during intercourse while taking drug and for condom is required to be used also by vasectomized men in order to prevent delivery of drug via seminal fluid.
* Patient is currently receiving (or has received within 4 weeks of baseline visit) VX-770/Ivacaftor.
* History of lung transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2012-07-31 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- United States (8):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Columbus, Ohio
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
- France (3):
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
- Germany (2):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Berlin
- Novartis Investigative Site, Dublin, Ireland
- Novartis Investigative Site, Bucharest, Romania
- United Kingdom (5):
  - Novartis Investigative Site, Livingston, West Lothian
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Mid Glamorgan

REFERENCES:
- [Derived] Kazani S, Rowlands DJ, Bottoli I, Milojevic J, Alcantara J, Jones I, Kulmatycki K, Machineni S, Mostovy L, Nicholls I, Nick JA, Rowe SM, Simmonds NJ, Vegesna R, Verheijen J, Danahay H, Gosling M, Ayalavajjala PS, Salman M, Strieter R. Safety and efficacy of the cystic fibrosis transmembrane conductance regulator potentiator icenticaftor (QBW251). J Cyst Fibros. 2021 Mar;20(2):250-256. doi: 10.1016/j.jcf.2020.11.002. Epub 2020 Dec 6. PMID 33293212
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=127

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For Cohort 6 continuing into the food effect part of the study the subjects remained on the same treatment assignment that was required during the fed state. Therefore no randomization f the subject occurred during the food effect arm. Only 5 of the 6 subjects went into the fed cohort.
Pre-assignment Details: In parts 1 and 2, participants (Healthy Volunteers) were randomized 3:1 to receive QBW251X or placebo. In part 3, participants (cystic fibrosis (CF) patients) were randomized 3:1 to receive QBW251X or placebo.
Groups:
- Part 1 Cohort 6: QBW251 (Fasting/Fed), Same Subjects: Single dose of QBW251 500 mg (fed). single dose with food for a preliminary assessment of the effect of food on the absorption of QBW251 in Healthy Volunteers. Each treatment period was comprised of a baseline period (Day -1), an inpatient dosing period (Days 1 to 3), three follow-up visits (Days 4, 5, and 8), and one end-of-treatment-period evaluation performed 14 days after the dose of study drug (Day 15).
Period: Part 1 and 2 (Healthy Volunteers)
Arm/Group | Part 1 Cohort 1: QBW251 | Part 1 Cohort 2: QBW251 | Part 1 Cohort 3: QBW251 | Part 1 Cohort 4: QBW251 | Part 1 Cohort 5: QBW251 | Part 1 Cohort 6: QBW251 (Fasting/Fed), Same Subjects | Part 1 Cohort 7: QBW251 | Part 1 Cohort 8: QBW251 | Part 1 Placebo | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251 | Part 2 Placebo | Part 3 Cohort 1: QBW251 | Part 3 Cohort 2: QBW251 | Part 3 Cohort 3: QBW251 | Part 3 Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 6 | 6 | 6 | 6 | 6 | 10 | 0 | 0 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 6 | 6 | 6 | 6 | 5 | 8 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 3 (Patients)
Arm/Group | Part 1 Cohort 1: QBW251 | Part 1 Cohort 2: QBW251 | Part 1 Cohort 3: QBW251 | Part 1 Cohort 4: QBW251 | Part 1 Cohort 5: QBW251 | Part 1 Cohort 6: QBW251 (Fasting/Fed), Same Subjects | Part 1 Cohort 7: QBW251 | Part 1 Cohort 8: QBW251 | Part 1 Placebo | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251 | Part 2 Placebo | Part 3 Cohort 1: QBW251 | Part 3 Cohort 2: QBW251 | Part 3 Cohort 3: QBW251 | Part 3 Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 12 | 19 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 12 | 19 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1 Cohort 6: QBW251 (Fastin / Fed), Same Subjects: Single dose of QBW251 500 mg (fed). single dose with food for a preliminary assessment of the effect of food on the absorption of QBW251 in Healthy Volunteers. Each treatment period was comprised of a baseline period (Day -1), an inpatient dosing period (Days 1 to 3), three follow-up visits (Days 4, 5, and 8), and one end-of-treatment-period evaluation performed 14 days after the dose of study drug (Day 15).
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1: QBW251 | Part 1 Cohort 2: QBW251 | Part 1 Cohort 3: QBW251 | Part 1 Cohort 4: QBW251 | Part 1 Cohort 6: QBW251 | Part 1 Cohort 6: QBW251 (Fastin / Fed), Same Subjects | Part 1 Cohort 7: QBW251 | Part 1 Cohort 8: QBW251 | Part 1 Placebo | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251 | Part 2 Placebo | Part 3 Cohort 1: QBW251 | Part 3 Cohort 2: QBW251 | Part 3 Cohort 3: QBW251 | Part 3 Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 12 | 19 | 12 | 153
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Part 1, HV (n= 64) | 36.3 (8.69) | 35 (14.25) | 43.5 (3.39) | 33.3 (9.61) | 44.2 (8.23) | 43.6 (9.07) | 28.2 (9.28) | 33.2 (9.47) | 30.3 (9.18) | NA (NA) — This row is for Part 1 HV | NA (NA) — This row is for Part 1 HV | NA (NA) — This row is for Part 1 HV | NA (NA) — This row is for Part 1 HV | NA (NA) — This row is for Part 1 HV | NA (NA) — This row is for Part 1 HV | NA (NA) — This row is for Part 1 HV | NA (NA) — This row is for Part 1 HV | NA (NA) — This row is for Part 1 HV | NA (NA) — This row is for Part 1 HV | 34.4 (9.92)
  Part 2, HV (n=40) | NA (NA) — This row is for Part 2 HV | NA (NA) — This row is for Part 2 HV | NA (NA) — This row is for Part 2 HV | NA (NA) — This row is for Part 2 HV | NA (NA) — This row is for Part 2 HV | NA (NA) — This row is for Part 2 HV | NA (NA) — This row is for Part 2 HV | NA (NA) — This row is for Part 2 HV | NA (NA) — This row is for Part 2 HV | 30.3 (5.13) | 30.5 (5.89) | 29.2 (11.62) | 31.7 (13.22) | 27.8 (5) | 29 (6.22) | NA (NA) — This row is for Part 2 HV | NA (NA) — This row is for Part 2 HV | NA (NA) — This row is for Part 2 HV | NA (NA) — This row is for Part 2 HV | 29.7 (7.82)
  Part 3, CF patients (n=49) | NA (NA) — This row is for Part 3 HV | NA (NA) — This row is for Part 3 HV | NA (NA) — This row is for Part 3 HV | NA (NA) — This row is for Part 3 HV | NA (NA) — This row is for Part 3 HV | NA (NA) — This row is for Part 3 HV | NA (NA) — This row is for Part 3 HV | NA (NA) — This row is for Part 3 HV | NA (NA) — This row is for Part 3 HV | NA (NA) — This row is for Part 3 HV | NA (NA) — This row is for Part 3 HV | NA (NA) — This row is for Part 3 HV | NA (NA) — This row is for Part 3 HV | NA (NA) — This row is for Part 3 HV | NA (NA) — This row is for Part 3 HV | 39.3 (5.47) | 32.7 (13.77) | 27 (5.44) | 27.9 (6.37) | 30.1 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 9 | 4 | 19
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 6 | 6 | 6 | 6 | 6 | 10 | 5 | 7 | 10 | 8 | 134

OUTCOME MEASURES:

1. Primary Outcome: Part 1 and 2:Number of Participants (Healthy Volunteers) With Reported Adverse Events Receiving QBW251
Description: All adverse events (in healthy volunteers) reported.
Time Frame: Day 1 to Day 36
Population: All treated subjects were included in the data analysis. Subjects were analyzed according to the study treatment(s) received.
Measure: Number; unit: Participants
Groups:
- Part 1 Cohort 1: QBW251: Single dose of QBW251 10 mg in Healthy Volunteers. Each treatment period was comprised of a baseline period (Day -1), an inpatient dosing period (Days 1 to 3), three follow-up visits (Days 4, 5, and 8), and one end-of-treatment-period evaluation performed 14 days after the dose of study drug (Day 15
Arm/Group | Part 1 Cohort 4: QBW251 | Part 1 Cohort 5: QBW251 | Part 1 Cohort 6: QBW251 | Part 1 Cohort 6: QBW251(Fed) | Part 1 Cohort 7: QBW251 | Part 1 Cohort 8: QBW251 | Part 1 Placebo | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251 | Part 2 Placebo | Part 1 Cohort 1: QBW251 | Part 1 Cohort 2: QBW251 | Part 1 Cohort 3: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 6 | 16 | 6 | 6 | 6 | 6 | 6 | 10 | 6 | 6 | 6
Participants
  Adverse events | 1 | 2 | 2 | 1 | 1 | 4 | 8 | 3 | 6 | 3 | 6 | 4 | 7 | 3 | 2 | 0
  Serious adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part 3: Change in Lung Clearance Index (LCI) From Baseline to Day 15
Description: Change in Lung Clearance Index (LCI) will be conducted according to international standards in cystic fibrosis patients. Lung clearance index (LCI) is a measure of ventilation inhomogeneity that is derived from a multiple-breath washout test, A reduction in mean change from baseline for LCI2.5 indicates improvement.
Time Frame: Baseline and Day 15
Population: Pharmacodynamics (PD) analysis set: All randomized patients were included in the PD analysis
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 3 Cohort 1: QBW251 | Part 3 Cohort 2: QBW251 | Part 3 Cohort 3: QBW251 | Part 3 Placebo
Number analyzed (Participants) | 5 | 11 | 17 | 11
Ratio | 0.27 (0.769) | -0.85 (1.798) | -0.13 (2.276) | 0.28 (1.959)

3. Primary Outcome: Part 3: Number of Participants (Patients) With Reported Adverse Events Receiving QBW251
Description: All adverse events and serious adverse events (in patients) reported.
Time Frame: Day 1 to Day 56
Population: Safety analysis set: All randomized patients were included in the safety analysis
Measure: Number; unit: Participants
Arm/Group | Part 3 Cohort 1: QBW251 | Part 3 Cohort 2: QBW251 | Part 3 Cohort 3: QBW251 | Part 3 Placebo
Number analyzed (Participants) | 6 | 12 | 19 | 12
Participants
  Adverse Events (AE) | 6 | 8 | 18 | 8
  Serious Adverse Events (SAE) | 1 | 1 | 1 | 0

4. Secondary Outcome: Part 3:Change in Forced Expiratory Volume in 1 Second (FEV1) at Day 15
Description: Forced Expiratory Volume in 1 second (FEV1) will be measured via spirometer according to international standards. Forced Expiratory Volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation
Time Frame: Baseline and Day 15
Population: Pharmacodynamics (PD) analysis set: All randomized patients were included in the PD analysis
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Part 3 Cohort 1: QBW251 | Part 3 Cohort 2: QBW251 | Part 3 Cohort 3: QBW251 | Part 3 Placebo
Number analyzed (Participants) | 5 | 11 | 16 | 12
Liters | 0.58 (2.476) | 5.99 (1.648) | -1.16 (1.059) | -1.46 (1.229)

5. Secondary Outcome: Part 3: Change in Cystic Fibrosis Questionnaire-Revised Reported Outcomes
Description: Change in Cystic Fibrosis Questionnaire data will be obtained from patient reported outcomes (CFQ-R PRO). Respiratory Domain, cores range from 0 to 100, with higher scores indicating better health, a change of 4 is considered clinically relevant
Time Frame: Baseline and Day 14
Population: Pharmacodynamics (PD) analysis set: All randomized patients were included in the PD analysis
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Part 3 Cohort 1: QBW251 | Part 3 Cohort 2: QBW251 | Part 3 Cohort 3: QBW251 | Part 3 Placebo
Number analyzed (Participants) | 5 | 11 | 19 | 12
Units on a scale | 16.06 (6.872) | 5.04 (4.617) | -2.62 (2.853) | -2.06 (4.415)

6. Secondary Outcome: Part 1: AUC0-t in Healthy Volunteers
Description: Pharmacokinetics of QBW251 in plasma: area under the plasma concentration versus time curve from time zero to time of last measurable concentration (AUC0-t). In part one of the study a single dose was administered and samples were collected up to 5 days. As a result the AUC0-t goes from Day 1 to Day 5 (for some lower doses QBW251 concentrations were not measured up to Day 5 as the concentrations were low due to the low dose administered)
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4 , 8 hr post-dose at Day 1; 24, 48, 72 and 96 hr post dose (i.e. Days 2-5)
Population: All subjects with at least one available valid (i.e. not flagged for exclusion) PK concentration measurement, who received study drug, and experienced no protocol deviations with relevant impact on PK data were included in the PK data analysis.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 1 Cohort 1: QBW251 | Part 1 Cohort 2: QBW251 | Part 1 Cohort 3: QBW251 | Part 1 Cohort 4: QBW251 | Part 1 Cohort 5: QBW251 | Part 1 Cohort 6: QBW251 | Part 1 Cohort 6: QBW251(Fed) | Part 1 Cohort 7: QBW251 | Part 1 Cohort 8: QBW251 | Part 1 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6 | 16
hr*ng/mL | 52.5 (28.1) | 73.7 (51.8) | 692 (389) | 1650 (907) | 5470 (1070) | 9450 (1740) | 7470 (2190) | 20200 (11500) | 35900 (9100) | NA (NA) — Not calculated

7. Secondary Outcome: Part 1: Maximum Concentration (Cmax) in Healthy Volunteers
Description: Pharmacokinetics of QBW251 in plasma: observed maximum plasma concentration following administration of QBW251. In this analysis Cmax will be reported using blood samples taken on Days 1- 5 are from healthy volunteers
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4 , 8 hr post-dose at Day 1; 24, 48, 72 and 96 hr post dose (i.e. Days 1 - 5)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Part 1 Cohort 1: QBW251 | Part 1 Cohort 2: QBW251 | Part 1 Cohort 3: QBW251 | Part 1 Cohort 4: QBW251 | Part 1 Cohort 5: QBW251 | Part 1 Cohort 6: QBW251 | Part 1 Cohort 6: QBW251(Fed) | Part 1 Cohort 7: QBW251 | Part 1 Cohort 8: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6
ug/L | 21.1 (11.9) | 24.7 (15.9) | 186 (82.3) | 459 (267) | 1110 (330) | 1910 (413) | 1090 (449) | 2680 (1000) | 4540 (930)

8. Secondary Outcome: Part 1: Time to Maximum Concentration (Tmax) in Healthy Volunteers
Description: Pharmacokinetics of QBW251 in plasma: time to reach the maximum concentration after administration of QBW251. In this analysis Tmax will be reported using blood samples taken on Days 1 - 5 from healthy volunteers. In this part of the study a single dose was administered and samples were collected up to 5 days. As a result the Tmax is one value as the concentration-time curve goes to Day 5 (for some lower does QBW251 concentrations were not measured up to Day 5 as the concentrations were low due to the low dose administered).
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4 , 8 hr post-dose at Day 1; 24, 48, 72 and 96 hr post dose (i.e. Days 1 - 5)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 1 Cohort 1: QBW251 | Part 1 Cohort 2: QBW251 | Part 1 Cohort 3: QBW251 | Part 1 Cohort 4: QBW251 | Part 1 Cohort 5: QBW251 | Part 1 Cohort 6: QBW251 | Part 1 Cohort 6: QBW251(Fed) | Part 1 Cohort 7: QBW251 | Part 1 Cohort 8: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6
hr | 0.756 (0.268) | 1.25 (0.612) | 1.33 (0.516) | 1.50 (0.548) | 1.50 (0.837) | 2.17 (1.17) | 3.40 (0.894) | 2.52 (0.850) | 1.83 (0.753)

9. Secondary Outcome: Part 1: T1/2 in Healthy Volunteers
Description: Pharmacokinetics of QBW251 in plasma: terminal elimination half-life. In this analysis T1/2 will be reported using blood samples taken on Days 1 - 5 from healthy volunteers. In part one of the study a single dose was administered and samples were collected up to 5 days. As a result the T1/2 goes from Day 1 to Day 5 (for some lower doses QBW251 concentrations were not measured up to Day 5 as the concentrations were low due to the low dose administered).
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4 , 8 hr post-dose at Day 1; 24, 48, 72 and 96 hr post dose (i.e. Days 1 - 5)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 1 Cohort 1: QBW251 | Part 1 Cohort 2: QBW251 | Part 1 Cohort 3: QBW251 | Part 1 Cohort 4: QBW251 | Part 1 Cohort 5: QBW251 | Part 1 Cohort 6: QBW251 | Part 1 Cohort 6: QBW251(Fed) | Part 1 Cohort 7: QBW251 | Part 1 Cohort 8: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6
hr | NA (NA) — There were not enough time points to calculated the T1/2 | NA (NA) — There were not enough time points to calculated the T1/2 | 10.3 (4.24) | 10.1 (3.35) | 12.0 (2.26) | 12.7 (1.99) | 15.6 (5.03) | 12.8 (3.85) | 10.7 (2.19)

10. Secondary Outcome: Part 1: AUCinf in Healthy Volunteers
Description: Pharmacokinetics of QBW251 in plasma: area under the plasma concentration time curve from time zero to infinity. In this analysis AUCinf will be reported using blood samples taken on Days 1 - 5 from healthy volunteers. In part one of the study a single dose was administered and samples were collected up to 5 days. As a result the AUCinf goes from Day 1 to Day 5 (for some lower doses QBW251 concentrations were not measured up to Day 5 as the concentrations were low due to the low dose administered)
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4 , 8 hr post-dose at Day 1; 24, 48, 72 and 96 hr post dose (i.e. Days 1 - 5)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 1 Cohort 1: QBW251 | Part 1 Cohort 2: QBW251 | Part 1 Cohort 3: QBW251 | Part 1 Cohort 4: QBW251 | Part 1 Cohort 5: QBW251 | Part 1 Cohort 6: QBW251 | Part 1 Cohort 6: QBW251(Fed) | Part 1 Cohort 7: QBW251 | Part 1 Cohort 8: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6
hr*ng/mL | NA (NA) — Not calculated due to insufficient data | NA (NA) — Not calculated due to insufficient data | 731 (387) | 1680 (903) | 5510 (1080) | 9480 (1740) | 7540 (2220) | 20300 (11500) | 36000 (9120)

11. Secondary Outcome: Part 1: CL/F in Healthy Volunteers
Description: Pharmacokinetics of QBW251 in plasma: apparent systemic clearance from plasma following extravascular administration. In this analysis CL/F will be reported using blood samples taken on Days 1 - 5 from healthy volunteers. In part one of the study a single dose was administered and samples were collected up to 5 days. As a result the CL/F goes from Day 1 to Day 5 (for some lower doses QBW251 concentrations were not measured up to Day 5 as the concentrations were low due to the low dose administered)
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4 , 8 hr post-dose at Day 1; 24, 48, 72 and 96 hr post dose (i.e. Days 1 - 5)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part 1 Cohort 1: QBW251 | Part 1 Cohort 2: QBW251 | Part 1 Cohort 3: QBW251 | Part 1 Cohort 4: QBW251 | Part 1 Cohort 5: QBW251 | Part 1 Cohort 6: QBW251 | Part 1 Cohort 6: QBW251(Fed) | Part 1 Cohort 7: QBW251 | Part 1 Cohort 8: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6
L/hr | NA (NA) — Not calculated due to insufficient data | NA (NA) — Not calculated due to insufficient data | 123 (49.0) | 114 (63.9) | 56.2 (11.0) | 54.5 (11.9) | 71.6 (22.6) | 45.9 (19.9) | 29.7 (9.00)

12. Secondary Outcome: Part 1: Vz/F in Healthy Volunteers
Description: Pharmacokinetics of QBW251 in plasma: apparent volume of distribution during the terminal elimination phase following extravascular administration. In this analysis Vz/F will be reported using blood samples taken on Days 1 - 5 from healthy volunteers.
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4 , 8 hr post-dose at Day 1; 24, 48, 72 and 96 hr post dose (i.e. Days 1 - 5)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part 1 Cohort 1: QBW251 | Part 1 Cohort 2: QBW251 | Part 1 Cohort 3: QBW251 | Part 1 Cohort 4: QBW251 | Part 1 Cohort 5: QBW251 | Part 1 Cohort 6: QBW251 | Part 1 Cohort 6: QBW251(Fed) | Part 1 Cohort 7: QBW251 | Part 1 Cohort 8: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 6
Liters | NA (NA) — Not calculated due to insufficient data | NA (NA) — Not calculated due to insufficient data | 1700 (772) | 1490 (622) | 957 (151) | 995 (235) | 1580 (587) | 827 (375) | 447 (112)

13. Secondary Outcome: Part 2: AUCtau in Healthy Volunteers
Description: Pharmacokinetics of QBW251 in plasma after multiple doses: the area under the plasma concentration-time curve from time zero to end of the dosing interval tau. In this analysis AUCtau will be reported. Samples taken on Days 1 and 14 from healthy volunteers
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4 , 8 hr post-dose at Day 1; 24, 48, 72 and 96 hr post dose Day 1 and 14; ( If B ID dosing, 12 hours samples will be pre-dosed)
Population: Pharmacokinetics analysis: All subjects with at least one available valid (i.e. not flagged for exclusion) PK concentration measurement, who received study drug, and experienced no protocol deviations with relevant impact on PK data were included in the PK data analysis
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hr*ng/mL
  Day1 | 1800 (794) | 6170 (1250) | 16100 (8170) | 7160 (1960) | 18800 (6360)
  Day 14 | 2060 (708) | 7620 (1470) | 28300 (5570) | 12100 (4930) | 80300 (56300)

14. Secondary Outcome: Part 2: Maximum Concentration (Cmax) in Healthy Volunteers
Description: Pharmacokinetics of QBW251 in plasma after multiple doses: observed maximum plasma concentration following QBW251 at steady state. In this analysis Cmax will be reported using blood samples taken on Days 1 and 14 from healthy volunteers.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ug/L
  Day 1 | 541 (338) | 1650 (343) | 2790 (1040) | 1650 (188) | 3720 (1530)
  Day 14 | 430 (145) | 1500 (442) | 3840 (868) | 2190 (769) | 9420 (4330)

15. Secondary Outcome: Part 2: Time to Maximum Concentration (Tmax) in Healthy Volunteers
Description: Pharmacokinetics of QBW251 in plasma after multiple doses: time to reach the maximum concentration after administration of QBW251. In this analysis Tmax will be reported using blood samples taken on Days 1 and 14 from healthy volunteers.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hr
  Day 1 | 1.67 (0.816) | 1.17 (0.408) | 2.33 (1.21) | 2.68 (0.813) | 3.67 (0.516)
  Day 2 | 2.17 (1.17) | 2.17 (0.408) | 2.33 (1.03) | 3.25 (1.41) | 3.80 (0.447)

16. Secondary Outcome: Part 2: AUC0-t
Description: Pharmacokinetics of QBW251 in plasma: area under the plasma concentration versus time curve from time zero to time of last measurable concentration. In this analysis AUC0-t will be reported using blood samples taken on Day 14 are from healthy volunteers.
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4 , 8 hr post-dose at Day 1; 24, 48, 72 and 96 hr post dose Day 14; ( If B ID dosing, 12 hours samples will be pre-dosed)
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251 | Part 2 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 14
hr*ng/mL | 2060 (708) | 7620 (1470) | 28300 (5570) | 12100 (4930) | 80300 (56300) | NA (NA) — Not calculated

17. Secondary Outcome: Part 2: Cav in Healthy Volunteers
Description: The average drug concentration in plasma during multiple dosing. In this analysis Cav will be reported using blood samples taken on Days 1 and 14 are from healthy volunteers.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ug/L | 85.8 (29.5) | 318 (61.1) | 1180 (232) | NA (NA) — Not calculated due to insufficient data | NA (NA) — Not calculated due to insufficient data

18. Secondary Outcome: Part 2: CL/F in Healthy Volunteers
Description: apparent systemic clearance from plasma following extravascular administration. In this analysis CL/F will be reported using blood samples taken on Day 14 from healthy volunteers.
Time Frame: as for outcome 16
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
L/hr | 80.8 (29.7) | 54.0 (9.40) | 27.5 (5.98) | NA (NA) — Not calculated due to insufficient data | NA (NA) — Not calculated due to insufficient data

19. Secondary Outcome: Part 2: Vz/F in Healthy Volunteers
Description: Apparent volume of distribution during the terminal elimination phase following extravascular administration. In this analysis Vz/F will be reported using blood samples taken on Day 14 from healthy volunteers.
Time Frame: as for outcome 16
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Liters | 1330 (550) | 1120 (395) | 608 (255) | NA (NA) — Not calculated due to insufficient data | NA (NA) — Not calculated due to insufficient data

20. Secondary Outcome: Part 2: Racc in Healthy Volunteers
Description: Accumulation ratio (Racc). In this analysis Racc will be reported using blood samples taken on Days 1 - 14 from healthy volunteers.
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4 , 8 hr post-dose at Day 1; 24, 48, 72 and 96 hr post dose Day 1 - 14; ( If B ID dosing, 12 hours samples will be pre-dosed)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
Ratio | 1.27 (0.425) | 1.25 (0.199) | 2.08 (0.913) | 1.66 (0.386) | 3.88 (2.07)

21. Secondary Outcome: Part 2: T1/2 in Healthy Volunteers
Description: terminal elimination half-life (T1/2). In this analysis T1/2 will be reported using blood samples taken on Day 14 from healthy volunteers.
Time Frame: as for outcome 16
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hr | 11.3 (1.44) | 14.1 (3.80) | 15.1 (4.40) | NA (NA) — Not calculated due to insufficient data | NA (NA) — Not calculated due to insufficient data

22. Secondary Outcome: Part 3: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of QBW251 in CF Patients
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4, 8 hr post-dose in Day 1, Day 14
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng × hr /mL
Arm/Group | Part 3 Cohort 1: QBW251 | Part 3 Cohort 2: QBW251 | Part 3 Cohort 3: QBW251
Number analyzed (Participants) | 6 | 12 | 19
ng × hr /mL
  Day 1 | 1110 (709) | 7530 (2480) | 6020 (2960)
  Day 14 | 1760 (943) | 18900 (6850) | NA (NA) — PK parameters were not calculated for Day 14 as blood samples were collected up to 2 hours post-dose.

23. Secondary Outcome: Part 3: Plasma Concentration at the Last Quantifiable Time Point (Clast) of QBW251 in CF Patients
Description: Blood samples were collected at timepoints prespecified in the study protocol. Tlast of QBW251 was the last time point when blood sample collected was quantifiable
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4, 8 hr post-dose in Day 1, Day2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 3 Cohort 1: QBW251 | Part 3 Cohort 2: QBW251 | Part 3 Cohort 3: QBW251
Number analyzed (Participants) | 6 | 12 | 19
ng/mL
  Day 1 | 42.3 (14.1) | 423 (275) | 653 (318)
  Day 14 | 86.4 (16.3) | 1570 (813) | NA (NA) — PK parameters were not calculated for Day 14 as blood samples were collected up to 2 hours post-dose

24. Secondary Outcome: Part 3: Maximum Concentration (Cmax) in CF Patients
Description: Observed maximum plasma concentration following administration of QBW251. In this analysis Cmax will be reported using blood samples taken on Day 1and day 14 from patients
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4, 8 hr post-dose in Day 1, Day 14
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 3 Cohort 1: QBW251 | Part 3 Cohort 2: QBW251 | Part 3 Cohort 3: QBW251
Number analyzed (Participants) | 6 | 12 | 19
ng/mL
  Day 1 | 419 (316) | 1950 (715) | 2380 (1240)
  Day 14 | 632 (438) | 4080 (1780) | NA (NA) — PK parameters were not calculated for Day 14 as blood samples were collected up to 2 hours post-dose

25. Secondary Outcome: Part 3: Tlast in CF Patients
Description: Blood samples were collected at timepoints prespecified in the study protocol. Tlast of QBW251 was the last time point when blood sample collected was quantifiable day 1 and day 14
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4, 8 hr post-dose in Day 1, Day 14
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 3 Cohort 1: QBW251 | Part 3 Cohort 2: QBW251 | Part 3 Cohort 3: QBW251
Number analyzed (Participants) | 6 | 12 | 19
hr
  Day 1 | 7.99 (0.0136) | 7.95 (0.149) | 5.80 (0.639)
  Day 14 | 7.97 (0.0667) | 7.96 (0.0554) | NA (NA) — PK parameters were not calculated for Day 14 as blood samples were collected up to 2 hours post-dose

26. Secondary Outcome: Part 3: Time to Maximum Concentration (Tmax)
Description: Pharmacokinetics of QBW251 in plasma after multiple doses: time to reach the maximum concentration after administration of QBW251. In this analysis Tmax will be reported using blood samples taken on Days 1 and 14 in patients
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4, 8 hr post-dose in Day 1, Day 14
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Part 3 Cohort 1: QBW251 | Part 3 Cohort 2: QBW251 | Part 3 Cohort 3: QBW251
Number analyzed (Participants) | 6 | 12 | 19
hr
  Day 1 | 3.17 (2.47) | 3.08 (1.68) | 3.18 (0.838)
  Day 14 | 1.82 (0.750) | 2.39 (0.973) | NA (NA) — PK parameters were not calculated for Day 14 as blood samples were collected up to 2 hours post-dose

27. Secondary Outcome: Part 2: Ae0-t in Healthy Volunteers
Description: Pharmacokinetics of QBW251 in urine: amount of drug excreted in urine from time zero until last measurable concentration. In this analysis Ae0-t will be reported using urine samples taken on Day 1 from healthy volunteers.
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4 , 8 hr post-dose at Day 1; 24, 48, 72 and 96 hr post dose Day 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251 | Part 2 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 5 | 14
L/hr | 2.36 (1.84) | 2.20 (1.26) | 1.21 (0.697) | 0.419 (0.271) | 0.140 (0.0936) | NA (NA) — Not calculated

28. Secondary Outcome: Part 2: CLr in Healthy Volunteers
Description: Pharmacokinetics of QBW251 in urine: renal clearance following drug administration. In this analysis CLr will be reported using urine samples taken on Day 1 from healthy volunteers.
Time Frame: Pre-dose (0 hr), 0.25, 0.5, 1, 2, 3, 4 , 8 hr post-dose at Day 1; 24, 48, 72 and 96 hr post dose Day 1; Day 14 was calculated as urine was only collected up to 12 hours on Day 1 thus CLr cannot be calculated.
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Part 2 Cohort 1: QBW251 | Part 2 Cohort 2: QBW251 | Part 2 Cohort 3: QBW251 | Part 2 Cohort 4: QBW251 | Part 2 Cohort 5: QBW251
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
L/hr | 2.36 (1.84) | 2.20 (1.26) | 1.21 (0.697) | 0.419 (0.271) | 0.140 (0.0936)

ADVERSE EVENTS:
Groups:
- Part 1 Placebo: Part 1 Placebo
- Part 1 QBW251 10mg: Part 1 QBW251 10mg
- Part 1 QBW251 25mg: Part 1 QBW251 25mg
- Part 1 QBW251 150mg: Part 1 QBW251 150mg
- Part 1 QBW251 300mg: Part 1 QBW251 300mg
- Part 1 QBW251 500mg: Part 1 QBW251 500mg
- Part 1 QBW251 500mg (Fed): Part 1 QBW251 500mg (fed)
- Part 1 QBW251 750mg: Part 1 QBW251 750mg
- Part 1 QBW251 1000mg: Part 1 QBW251 1000mg
- Part 2 Placebo: Part 2 Placebo
- Part 2 QBW251 150mg: Part 2 QBW251 150mg
- Part 2 QBW251 400mg: Part 2 QBW251 400mg
- Part 2 QBW251 750mg: Part 2 QBW251 750mg
- Part 2 QBW251 450mg BID: Part 2 QBW251 450mg BID
- Part 2 QBW251 750mg BID: Part 2 QBW251 750mg BID
- Part 3 Placebo C1/C2/C3: Part 3 Placebo C1/C2/C3
- Part 3 QBW251 150mg BID C1: Part 3 QBW251 150mg BID C1
- Part 3 QBW251 450mg BID C2: Part 3 QBW251 450mg BID C2
- Part 3 QBW251 450mg BID C3: Part 3 QBW251 450mg BID C3
Arm/Group | Part 1 Placebo | Part 1 QBW251 10mg | Part 1 QBW251 25mg | Part 1 QBW251 150mg | Part 1 QBW251 300mg | Part 1 QBW251 500mg | Part 1 QBW251 500mg (Fed) | Part 1 QBW251 750mg | Part 1 QBW251 1000mg | Part 2 Placebo | Part 2 QBW251 150mg | Part 2 QBW251 400mg | Part 2 QBW251 750mg | Part 2 QBW251 450mg BID | Part 2 QBW251 750mg BID | Part 3 Placebo C1/C2/C3 | Part 3 QBW251 150mg BID C1 | Part 3 QBW251 450mg BID C2 | Part 3 QBW251 450mg BID C3
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 1/6 | 1/12 | 1/19
Other Adverse Events (participants affected / at risk) | 8/16 | 3/6 | 2/6 | 1/6 | 2/6 | 2/6 | 1/5 | 1/6 | 4/6 | 7/10 | 3/6 | 6/6 | 3/6 | 6/6 | 4/6 | 8/12 | 5/6 | 8/12 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Placebo (N=16) | Part 1 QBW251 10mg (N=6) | Part 1 QBW251 25mg (N=6) | Part 1 QBW251 150mg (N=6) | Part 1 QBW251 300mg (N=6) | Part 1 QBW251 500mg (N=6) | Part 1 QBW251 500mg (Fed) (N=5) | Part 1 QBW251 750mg (N=6) | Part 1 QBW251 1000mg (N=6) | Part 2 Placebo (N=10) | Part 2 QBW251 150mg (N=6) | Part 2 QBW251 400mg (N=6) | Part 2 QBW251 750mg (N=6) | Part 2 QBW251 450mg BID (N=6) | Part 2 QBW251 750mg BID (N=6) | Part 3 Placebo C1/C2/C3 (N=12) | Part 3 QBW251 150mg BID C1 (N=6) | Part 3 QBW251 450mg BID C2 (N=12) | Part 3 QBW251 450mg BID C3 (N=19)
INFECTIVE PULMONARY EXACERBATION OF CYSTIC FIBROSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Placebo (N=16) | Part 1 QBW251 10mg (N=6) | Part 1 QBW251 25mg (N=6) | Part 1 QBW251 150mg (N=6) | Part 1 QBW251 300mg (N=6) | Part 1 QBW251 500mg (N=6) | Part 1 QBW251 500mg (Fed) (N=5) | Part 1 QBW251 750mg (N=6) | Part 1 QBW251 1000mg (N=6) | Part 2 Placebo (N=10) | Part 2 QBW251 150mg (N=6) | Part 2 QBW251 400mg (N=6) | Part 2 QBW251 750mg (N=6) | Part 2 QBW251 450mg BID (N=6) | Part 2 QBW251 750mg BID (N=6) | Part 3 Placebo C1/C2/C3 (N=12) | Part 3 QBW251 150mg BID C1 (N=6) | Part 3 QBW251 450mg BID C2 (N=12) | Part 3 QBW251 450mg BID C3 (N=19)
PALPITATIONS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
ICHTHYOSIS (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
EAR DISCOMFORT (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TINNITUS (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
FAECES DISCOLOURED (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
FLATULENCE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
GINGIVAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4 | 2
SALIVA ALTERED (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SALIVARY GLAND PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
ASTHENIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
CHEST DISCOMFORT (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FATIGUE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
PERIPHERAL SWELLING (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PYREXIA (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
SENSATION OF FOREIGN BODY (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
THIRST (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
VESSEL PUNCTURE SITE BRUISE (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BRONCHOPULMONARY ASPERGILLOSIS ALLERGIC (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
FOLLICULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INFECTIVE PULMONARY EXACERBATION OF CYSTIC FIBROSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ORAL HERPES (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PHARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SKIN WOUND (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ADENOVIRUS TEST POSITIVE (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BLOOD POTASSIUM DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BREATH SOUNDS ABNORMAL (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CORONAVIRUS TEST POSITIVE (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
BALANCE DISORDER (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
HEADACHE (Nervous system disorders) | 2 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 4 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 3 | 4
HYPERAESTHESIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
TREMOR (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
AGITATION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
INSOMNIA (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
STRESS (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CHROMATURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
GLYCOSURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PROTEINURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 2 | 1 | 1 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
PAINFUL RESPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SPUTUM INCREASED (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 5
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
TONSILLAR DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
HEAT RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HOT FLUSH (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.